CLINICAL TRIAL: NCT03146598
Title: Use and Tolerability of a Side Pole Static Ankle Foot Orthosis in Children With Neurological Disorders
Brief Title: Side Pole Static Ankle Foot Orthosis in Children With Neurological Disorders
Acronym: SPS-AFO
Status: Completed | Type: Observational
Sponsor: BERTHILLIER Julien (Other)
Responsible Party: Sponsor-Investigator, BERTHILLIER Julien, Project manager, Hospices Civils de Lyon
Organization: Hospices Civils de Lyon (Other)
Other Study IDs: 2015-68
Record Dates: First submitted 2017-05-02; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Neurological Disorder
Keywords: Foot deformity; Orthopaedic management; prevention; side pole static ankle foot orthosis
MeSH Terms: conditions — Nervous System Diseases; Foot Deformities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention as it is a observational study — No intervention as it is a observational study

SUMMARY:
Transverse-plane foot deformities are a frequently encountered issue in children with neurological disorders. They are the source of many symptoms, such as pain and walking difficulties, making their prevention very important. It is thus important to prevent the occurrence of transverse-plane foot deformities and limit their development regarding the high risk of morbidity. In order to prevent such deformities, in the department of pediatric physical medicine and rehabilitation department of Lyon, since 2001 the investigator use a side pole static ankle foot orthosis (SPS AFO) in children with a neurological disorder predisposing such deformities. The aim of the study this study is to describe the use, tolerability and potential side effects of this orthosis in children with neurological disorders from the investigator's department

ELIGIBILITY:
Inclusion Criteria:

* regularly follow-up in the department of physical medicine and pediatric rehabilitation L'Escale (Lyon, France)
* presenting at least unilateral transverse-plane foot deformity within the context of a neurological disorder
* having a first prescription of SPS AFO between December 2001 and December 2011.

Exclusion Criteria:

* None

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patient from the department of physical medicine and pediatric rehabilitation L'Escale (Lyon, France)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2012-01-01 (Actual); Study Completion 2012-01-01 (Actual)

PRIMARY OUTCOMES:
Duration of the SPS AFO wearing | At 3 months after SPS AFO implementation
  Duration of the SPS AFO wearing

SECONDARY OUTCOMES:
Frequency of the SPS AFO wearing | At 3 months after SPS AFO implementation
  Frequency of the SPS AFO wearing
Duration of the SPS AFO wearing | At 1 year after SPS AFO implementation
  Duration of the SPS AFO wearing
Frequency of the SPS AFO wearing | At 1 year after SPS AFO implementation
  Frequency of the SPS AFO wearing
Duration of the SPS AFO wearing | at 2 year after SPS AFO implementation
  Duration of the SPS AFO wearing
Frequency of the SPS AFO wearing | at 2 year after SPS AFO implementation
  Frequency of the SPS AFO wearing
Duration of the SPS AFO wearing | At 4 years after SPS AFO implementation
  Duration of the SPS AFO wearing
Frequency of the SPS AFO wearing | At 4 years after SPS AFO implementation
  Frequency of the SPS AFO wearing

IPD SHARING:
Plan to Share IPD: No